CLINICAL TRIAL: NCT03203759
Title: Hospital-Level Care at Home for Acutely Ill Adults: A Randomized Controlled Trial
Brief Title: Hospital-Level Care at Home for Acutely Ill Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Vital Connect (Unknown); Smiths Medical (Unknown)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P001337
Record Dates: First submitted 2017-06-05; First posted 2017-06-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Infection; Heart Failure; COPD; Asthma; Gout Flare; Chronic Kidney Diseases; Hypertensive Urgency; Atrial Fibrillation Rapid; Anticoagulants; Increased
MeSH Terms: conditions — Infections; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma; Renal Insufficiency, Chronic; Hypertensive Crisis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient hospitalization (Active Comparator): Control / usual care arm. Patients are admitted per usual to an inpatient service. Patients' medical records will be closely monitored. Patients will wear a vital sign and activity monitor whose data is used only retrospectively. On discharge and 30 days after discharge, they will be interviewed regarding their hospitalization and health.
  Interventions: Other: Traditional inpatient hospitalization
- Home hospitalization (Experimental): Intervention arm. Patients will return home after triage, diagnosis, and the beginning of treatment in the emergency department with a set of specialized patient-tailored services (listed above). On discharge and 30 days after discharge, they will be interviewed regarding their hospitalization and health.
  Interventions: Other: Home hospitalization

INTERVENTIONS:
Other: Home hospitalization — See above
  Arms: Home hospitalization
Other: Traditional inpatient hospitalization — See above
  Arms: Inpatient hospitalization

SUMMARY:
The investigators propose a home hospital model of care that substitutes for treatment in an acute care hospital. Limited studies of the home hospital model have demonstrated that a sizeable proportion of acute care can be delivered in the home with equal quality and safety, reduced cost, and improved patient experience.

DETAILED DESCRIPTION:
Hospitals are the standard of care for acute illness in the United States, but hospital care is expensive and often unsafe, especially for older individuals. While admitted, 20% suffer delirium, over 5% contract hospital-acquired infections, and most lose functional status that is never regained. Timely access to inpatient care is poor: many hospital wards are typically over 100% capacity, and emergency department waits can be protracted. Moreover, hospital care is increasingly costly: many internal medicine admissions have a negative margin (i.e., expenditures exceed hospital revenues) and incur patient debt.

The investigators propose a home hospital model of care that substitutes for treatment in an acute care hospital. Studies of the home hospital model have demonstrated that a sizeable proportion of acute care can be delivered in the home with equal quality and safety, 20% reduced cost, and 20% improved patient experience. While this is the standard of care in several developed countries, only 2 non-randomized demonstration projects have been conducted in the United States, each with highly local needs. Taken together, home hospital evidence is promising but falls short due to non-robust experimental design, failure to implement modern medical technology, and poor enlistment of community support.

The home hospital module offers most of the same medical components that are standard of care in an acute care hospital. The typical staff (medical doctor [MD], registered nurse [RN], case manager), diagnostics (blood tests, vital signs, telemetry, x-ray, and ultrasound), intravenous therapy, and oxygen/nebulizer therapy will all be available for home hospital. Optional deployment of food services, home health aide, physical therapist, occupational therapist, and social worker will be tailored to patient need. Home hospital improves upon the components of a typical ward's standard of care in several ways:

Point of care blood diagnostics (results at the bedside in <5 minutes); Minimally invasive continuous vital signs, telemetry, activity tracking, and sleep tracking; Automated alerting of MDs by mobile phone for any worrisome vital sign patterns; On-demand 24/7 clinician video visits; 4 to 1 patient to attending MD ratio, compared to typical 16 to 1; Ambulatory/portable infusion pumps that can be worn on the hip; Optional access to a personal home health aide.

Should a matter be emergent (that is, requiring in-person assistance in less than 20 minutes), then 9-1-1 will be called and the patient will be returned to the hospital immediately. In previous iterations of home hospital this happens in about 2% of patients.

Clinical parameters measured will be at the discretion of the physician and nurse, who treat the participant following evidence-based practice guidelines, just as in the usual care setting. In addition, the investigators will be tracking a wide variety of measures of quality and safety, including some measures tailored to each primary diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Resides within either a 5-mile or 20 minute driving radius of emergency department
* Has capacity to consent to study OR can assent to study and has proxy who can consent
* >= 18 years-old
* Can identify a potential caregiver who agrees to stay with patient for first 24 hours of admission. Caregiver must be competent to call care team if a problem is evident to her/him. After 24 hours, this caregiver should be available for as-needed spot checks on the patient. This criterion may be waived for highly competent patients at the patient and clinician's discretion.
* Primary or possible diagnosis of cellulitis, heart failure, complicated urinary tract infection, pneumonia, COPD/asthma, other infection, chronic kidney disease, malignant pain, diabetes and its complications, gout flare, hypertensive urgency, previously diagnosed atrial fibrillation with rapid ventricular response, anticoagulation needs, or a patient who desires only medical management that requires inpatient admission, as determined by the emergency room team.

Exclusion Criteria:

* Undomiciled
* No working heat (October-April), no working air conditioning if forecast > 80°F (June-September), or no running water
* On methadone requiring daily pickup of medication
* In police custody
* Resides in facility that provides on-site medical care (e.g., skilled nursing facility)
* Domestic violence screen positive
* Acute delirium, as determined by the Confusion Assessment Method
* Cannot establish peripheral access in emergency department (or access requires ultrasound guidance)
* Secondary condition: end-stage renal disease, acute myocardial infarction, acute cerebral vascular accident, acute hemorrhage
* Primary diagnosis requires multiple or routine administrations of intravenous narcotics for pain control
* Cannot independently ambulate to bedside commode
* As deemed by on-call medical doctor, patient likely to require any of the following procedures: computed tomography, magnetic resonance imaging, endoscopic procedure, blood transfusion, cardiac stress test, or surgery
* High risk for clinical deterioration
* Home hospital census is full (maximum 5 patients at any time)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-02-17 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Total direct cost of hospitalization, $ | From date of admission to date of discharge, an expected average of 4 days

SECONDARY OUTCOMES:
Direct margin, $ | From date of admission to date of discharge, an expected average of 4 days
  Direct margin from total cost of hospitalization
Direct margin, modeled with backfill | From date of admission to date of discharge, an expected average of 4 days
  Backfill uses a model that estimates the cost of patients who take the place of home hospital patients
Total cost, 30-day post discharge | Day of admission to 30-days post-discharge
Length of stay, days | From date of admission to date of discharge, an expected average of 4 days
Imaging, # | From date of admission to date of discharge, an expected average of 4 days
  Count of any diagnostic imaging (for example, x-ray, computed tomography, magnetic resonance, ultrasound, and nuclear imaging) that occurred through the course of the hospitalization.
Lab orders, # | From date of admission to date of discharge, an expected average of 4 days
  Count of any lab order (for example, basic metabolic panel, complete blood count, hepatic function panel) that occurred through the course of the hospitalization.
All-cause readmission(s) after index, # | Day of discharge to 30 days later
All-cause readmission(s) after index, y/n | Day of discharge to 30 days later
Unplanned readmission(s) after index, # | Day of discharge to 30 days later
Unplanned readmission(s) after index, y/n | Day of discharge to 30 days later
Emergency Department observation stay(s) after index hospitalization, # | Day of discharge to 30 days later
Emergency Department observation stay(s) after index hospitalization, y/n | Day of discharge to 30 days later
Emergency Department visit(s) after index hospitalization, # | Day of discharge to 30 days later
Emergency Department visit(s) after index hospitalization, y/n | Day of discharge to 30 days later
Delirium, y/n | From date of admission to date of discharge, an expected average of 4 days
Transfer back to hospital, y/n | From date of admission to date of discharge, an expected average of 4 days
  Intervention arm only
Hours of sleep per day, # | From date of admission to date of discharge, an expected average of 4 days
Hours of activity per day, # | From date of admission to date of discharge, an expected average of 4 days
Hours of sitting upright per day, # | From date of admission to date of discharge, an expected average of 4 days
Steps per day, # | From date of admission to date of discharge, an expected average of 4 days
EuroQol -5D-5L, composite score | At admission, at discharge (the day the patient leaves the hospital environment), and at 30 days after discharge
Short Form 1 | 30 days prior to admission (asked on day of admission), at admission, at discharge (the day the patient leaves the hospital environment), and at 30 days after discharge
  1-5 Likert scale
Activities of daily living, score | 30 days prior to admission (asked on day of admission), at admission, at discharge (the day the patient leaves the hospital environment), and at 30 days after discharge
Instrumental activities of daily living, score | 30 days prior to admission (asked on day of admission), at admission, at discharge (the day the patient leaves the hospital environment), and at 30 days after discharge
3-item Care Transition Measure, score | 30 days after discharge
Picker Experience Questionnaire, score | 30 days after discharge
Global satisfaction with care, score | 30 days after discharge
Qualitative interview | 30 days after discharge

OTHER OUTCOMES:
Total reimbursement, 30-day post discharge | Day of admission to 30-days post-discharge
  Exploratory
Intravenous medications, days | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Intravenous fluids, days | From date of admission to date of discharge, an expected average of 4 days
  Exploratory; the number of days intravenous fluids (for example, normal saline) were received by the patient.
Intravenous diuretics, days | From date of admission to date of discharge, an expected average of 4 days
  Exploratory; the number of days intravenous diuretics (for example, furosemide) were received by the patient.
Intravenous antibiotics, days | From date of admission to date of discharge, an expected average of 4 days
  Exploratory; the number of days intravenous antibiotics (for example, ceftriaxone) were received by the patient.
Supplemental oxygen required, days | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Nebulizer treatment, days | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Medical Doctor sessions, # notes | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Consultant sessions, # notes | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Physical therapy/occupational therapy sessions, # notes | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Primary care provider follow-up within 14 days, y/n | Day of discharge to 14 days later
  Exploratory
Skilled nursing facility utilization, days | Day of discharge to 30 days later
  Exploratory; the number of days a patient spent in a skilled nursing facility.
Home health utilization, days | Day of discharge to 30 days later
  Exploratory
Fall, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Hospital-acquired deep vein thrombosis or pulmonary embolism, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Hospital-acquired pressure ulcer, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Hospital-acquired thrombophlebitis at peripheral IV site, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Hospital-acquired catheter-associated urinary tract infection, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Hospital-acquired Clostridium difficile infection, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Hospital-acquired methicillin resistant staphylococcus aureus infection, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
All-cause mortality, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Unplanned mortality, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Post-discharge all-cause mortality, y/n | Day of discharge to 30 days later
  Exploratory
Post-discharge unplanned mortality, y/n | Day of discharge to 30 days later
  Exploratory
New arrhythmia, y/n | From date of admission to date of discharge, an expected average of 4 days
  Heart failure patients only; Exploratory
Hypokalemia, y/n | From date of admission to date of discharge, an expected average of 4 days
  Heart failure patients only; Exploratory
Acute Kidney Injury, y/n | From date of admission to date of discharge, an expected average of 4 days
  Heart failure patients only; Exploratory
Mean Likert scale pain score, 0-10 | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Hours of sleep per night, # | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Hours of activity per night, # | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Hours of sitting upright per night, # | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Pneumococcal vaccination if appropriate, y/n | From date of admission to date of discharge, an expected average of 4 days
  Pneumonia patients only; Exploratory
Influenza vaccination if appropriate, y/n | From date of admission to date of discharge, an expected average of 4 days
  Pneumonia patients only; Exploratory
Smoking cessation counseling if appropriate, y/n | From date of admission to date of discharge, an expected average of 4 days
  Pneumonia and heart failure patients only; Exploratory
Evaluation of ejection fraction as assessed by echocardiogram or other appropriate study, scheduled or completed, if not done within 1 year; y/n | From date of admission to date of discharge, an expected average of 4 days
  Heart failure patients only; Exploratory; Whether or not an appropriate study occurred and/or was scheduled if not done within 1 year; appropriate studies include cardiac magnetic resonance imaging, radionuclide ventriculography, single photon emission computed tomography myocardial perfusion imaging, or left ventriculography
Angiotensin converting enzyme inhibitor or angiotensin receptor blocker for heart failure with reduced ejection fraction (ejection fraction < 40%), y/n | From date of admission to date of discharge, an expected average of 4 days
  Heart failure patients only; Exploratory
Beta blocker for heart failure with reduced ejection fraction (ejection fraction < 40%), y/n | From date of admission to date of discharge, an expected average of 4 days
  Heart failure patients only; Exploratory
Aldosterone antagonist for heart failure with reduced ejection fraction (ejection fraction < 40%), y/n | From date of admission to date of discharge, an expected average of 4 days
  Heart failure patients only; Exploratory
Lipid lowering for coronary artery disease, peripheral vascular disease, cerebrovascular accident, or diabetes, y/n | From date of admission to date of discharge, an expected average of 4 days
  Heart failure patients only; Exploratory
Smoking status post-discharge; current/never/quit | From date of admission to date of discharge, an expected average of 4 days
  Heart failure and pneumonia patients only; Exploratory; Self-report of smoking status: current/never/quit.
Use of inappropriate medications in the elderly, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory; using Screening Tool of Older Persons' potentially inappropriate Prescriptions (STOPP) and Beers criteria
Use of Foley catheter, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
Use of restraints, y/n | From date of admission to date of discharge, an expected average of 4 days
  Exploratory
>3 medications added to medication list, y/n | Date of discharge, an expected average of 4 days after the date of admission
  Exploratory; comparison made between preadmission and discharge medication list
Patient health questionnaire-2, score | At admission, at discharge (an expected average of 4 days after the date of admission), and at 30 days after discharge
  Exploratory
Patient-Reported Outcomes Measurement Information System Emotional Support Short Form 4a, score | At admission, at discharge (an expected average of 4 days after the date of admission), and at 30 days after discharge
  Exploratory
Days at home since discharge | 30 days after discharge
  Exploratory
Walk around ward/home, y/n | Date of discharge, an expected average of 4 days after the date of admission
  Exploratory
Get to (non-commode) bathroom, y/n | Date of discharge, an expected average of 4 days after the date of admission
  Exploratory
Walk 1 flight of stairs, y/n | Date of discharge, an expected average of 4 days after the date of admission
  Exploratory
Visit with friends/family, y/n | Date of discharge, an expected average of 4 days after the date of admission
  Exploratory
Walk outside around my home, y/n | Date of discharge, an expected average of 4 days after the date of admission
  Exploratory
Go shopping, y/n | Date of discharge, an expected average of 4 days after the date of admission
  Exploratory
Time from admission decision to assessment by research assistant, minutes | On the first day of admission, a maximum 24 hour period
  Exploratory
Time from research assistant assessment to emergency department dismissal, minutes | On the first day of admission, a maximum 24 hour period
  Exploratory
Time from arrival home or to floor and medical doctor evaluation, minutes | On the first day of admission, a maximum 24 hour period
  Exploratory
Time from arrival home or to floor and registered nurse evaluation, minutes | On the first day of admission, a maximum 24 hour period
  Exploratory
Mean registered nurse to patient ratio | From date of admission to date of discharge, an expected average of 4 days
  Exploratory, intervention arm only
Total registered nurse visits, # | From date of admission to date of discharge, an expected average of 4 days
  Exploratory, intervention arm only
Total "on call" medical doctor interactions (video or phone), # | From date of admission to date of discharge, an expected average of 4 days
  Exploratory, intervention arm only
Total "on call" medical doctor in-person visits, # | From date of admission to date of discharge, an expected average of 4 days
  Exploratory, intervention arm only
Duration of 1st registered nurse visit, minutes | On the first day of admission, a maximum 24 hour period
  Exploratory, intervention arm only
Mean duration of subsequent registered nurse visit, minutes | From date of admission to date of discharge, an expected average of 4 days
  Exploratory, intervention arm only

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Schnipper, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leff B, Burton L, Mader SL, Naughton B, Burl J, Inouye SK, Greenough WB 3rd, Guido S, Langston C, Frick KD, Steinwachs D, Burton JR. Hospital at home: feasibility and outcomes of a program to provide hospital-level care at home for acutely ill older patients. Ann Intern Med. 2005 Dec 6;143(11):798-808. doi: 10.7326/0003-4819-143-11-200512060-00008. PMID 16330791
- [Background] Cryer L, Shannon SB, Van Amsterdam M, Leff B. Costs for 'hospital at home' patients were 19 percent lower, with equal or better outcomes compared to similar inpatients. Health Aff (Millwood). 2012 Jun;31(6):1237-43. doi: 10.1377/hlthaff.2011.1132. PMID 22665835
- [Background] Hung WW, Ross JS, Farber J, Siu AL. Evaluation of the Mobile Acute Care of the Elderly (MACE) service. JAMA Intern Med. 2013 Jun 10;173(11):990-6. doi: 10.1001/jamainternmed.2013.478. PMID 23608775
- [Background] Fong TG, Tulebaev SR, Inouye SK. Delirium in elderly adults: diagnosis, prevention and treatment. Nat Rev Neurol. 2009 Apr;5(4):210-20. doi: 10.1038/nrneurol.2009.24. PMID 19347026
- [Background] Counsell SR, Holder CM, Liebenauer LL, Palmer RM, Fortinsky RH, Kresevic DM, Quinn LM, Allen KR, Covinsky KE, Landefeld CS. Effects of a multicomponent intervention on functional outcomes and process of care in hospitalized older patients: a randomized controlled trial of Acute Care for Elders (ACE) in a community hospital. J Am Geriatr Soc. 2000 Dec;48(12):1572-81. doi: 10.1111/j.1532-5415.2000.tb03866.x. PMID 11129745
- [Background] Montalto M. The 500-bed hospital that isn't there: the Victorian Department of Health review of the Hospital in the Home program. Med J Aust. 2010 Nov 15;193(10):598-601. doi: 10.5694/j.1326-5377.2010.tb04070.x. PMID 21077817
- [Derived] Levine DM, Paz M, Burke K, Schnipper JL. Predictors and Reasons Why Patients Decline to Participate in Home Hospital: a Mixed Methods Analysis of a Randomized Controlled Trial. J Gen Intern Med. 2022 Feb;37(2):327-331. doi: 10.1007/s11606-021-06833-2. Epub 2021 May 5. PMID 33954888
- [Derived] Levine DM, Pian J, Mahendrakumar K, Patel A, Saenz A, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: a Qualitative Evaluation of a Randomized Controlled Trial. J Gen Intern Med. 2021 Jul;36(7):1965-1973. doi: 10.1007/s11606-020-06416-7. Epub 2021 Jan 21. PMID 33479931
- [Derived] Levine DM, Ouchi K, Blanchfield B, Saenz A, Burke K, Paz M, Diamond K, Pu CT, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: A Randomized Controlled Trial. Ann Intern Med. 2020 Jan 21;172(2):77-85. doi: 10.7326/M19-0600. Epub 2019 Dec 17. PMID 31842232